CLINICAL TRIAL: NCT05915364
Title: MAgna GraecIa Evaluation of Comorbidities in Patients With Heart Failure STUDY (MAGIC-HF STUDY): Observational Study on Physiopathological, Diagnostic, Therapeutic, and Predictive Aspects of Heart Failure and Associated Comorbidities
Brief Title: MAgna GraecIa Evaluation of Comorbidities in Patients With Heart Failure STUDY
Acronym: MAGIC-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Angela Sciacqua, Associate Professor, University of Catanzaro
Other Study IDs: 304.2022
Record Dates: First submitted 2023-05-10; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure
Keywords: heart failure; biomarkers; cardiovascular complications; Prevention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum samples, Blood samples, Lymphocytes preparations, Stools samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HF patients: Adult subjects with all forms of HF will be recruited

SUMMARY:
The MAGIC-HF STUDY project (MAgna GraecIa evaluation of Comorbidities in patients with Heart Failure STUDY), is an observational prevalence and incidence study focusing on the role that risk factors, various comorbidities, and their treatment may have on CV and non-CV outcomes in patients with all forms of HF. It also aim to assess whether comorbidities and their treatment may be predictors of response to pharmacological and non-drug treatment of HF.

DETAILED DESCRIPTION:
Adult subjects with all forms of HF (HFrEF, HFmrEf, HEpEF) with at least one comorbidity who are referred to the Heart Failure Outpatient Clinic of the AOU "Mater Domini" Geriatrics Unit in Catanzaro will be recruited.

Initially, patients will be evaluated at baseline and followed-up for a minimum of six-month.

All patients will be subjected to clinical, instrumental and laboratory examinations, including medical history data collection and complete anthropometric assessment . Plasma and serum samples will be collected at recruitment and at the six-months follow-up visit. Stool samples will also be obtained and stored at -80C for the omics studies.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent obtained before performing any procedure
* Age>18 years old
* Confirmed diagnosis of HFrEF, HFmrEF, HFpEF with clinical stability for at least 4 weeks
* Presence of at least one of the following comorbidities:
* Atrial fibrillation
* Peripheral arteriopathy
* Hypertension
* Chronic ischemic heart disease
* Diabetes mellitus type 2 or insulin resistance
* Hepatopathy
* Obesity
* Cancer
* Sleep apnea syndrome
* Chronic kidney disease
* Iron deficiency
* Cognitive Decline or Depression
* Sarcopenia
* Dysthyroidisms
* Hypovitaminosis D
* Hyperuricemia

Exclusion Criteria:

* Liver cirrhosis Child-Pugh C
* Severe chronic renal failure defined by an estimated glomerular filtration rate (eGFR) value < 15 ml/min/1.73 m2 according to CKD-EPI
* Suspected alcohol or drug abuse
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients referred to the outpatient heart failure clinic of the Geriatrics Units of Mater Domini Hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of cardiac parameters | 6 months
  Echocardiographic evaluation of the left ventricular global system, left ventricular ejection fraction, left atrial diameter, cardiac output, cardiac index, right ventricular global function by Color-Doppler echocardiogram (Vivid E95, GE Healthcare, Horten, Norway)
Spekle-tracking Imaging | 6 months
  A 2D speckle tracking analysis was retrospectively performed using vendor-specific 2D speckle tracking software (EchoPAC PC, version 113.0.5, GE Healthcare, Horten, Norway). Manual tracings of the endocardial border during end-systole in three apical views was performed to evaluate GLS.
  echocardiogram (Vivid E95, GE Healthcare, Horten, Norway)
Determination of intimal media thickness | 6 months
  Determination of intimal media thickness by high-resolution ultrasonography of common carotid arteries
MiniMental State examination | 6 months
  Geriatric multidimensional assessment for the evaluation of MiniMental State examination (MMSE), in patients over 65 years old (range values 0-30 score).
Geriatric depression scale | 6 months
  Geriatric multidimensional assessment for the evaluation of Geriatric depression scale (GDS) in patients over 65 years old. The short form (GDS-S) consists of 15 items. Of the 15 elements, 10 indicate the presence of depression when responding positively, while the other five are indicative of depression when responding negatively, moreover > 5 points suggest depression and require follow-up evaluation, ≥ 10 points almost always indicates depression.
Montreal Cognitive Assessment | 6 months
  Geriatric multidimensional assessment for the evaluation of Montreal Cognitive Assessment (MoCA) in patients over 65 years old. This one-page 30-point test can be administered to the patient in at last 10 min. Cut-off score 26 points.
Evaluation of autonomy in daily activities | 6 months
  Geriatric multidimensional assessment for the evaluation of autonomy in daily activities living (ADL) in patients over 65 years old. The score ranges from 0/6 (maximum dependence) to 6/6 (maximum autonomy).
Autonomy in instrumental activities of daily living | 6 months
  Geriatric multidimensional assessment for the evaluation of autonomy in instrumental activities of daily living (IADL) in patients over 65 years old. Range values 0-8 points.
Short Performance Physical battery | 6 months
  Geriatric multidimensional assessment for the evaluation of Short Performance Physical battery (SPPB) in patients over 65 years old. The total score of the scale has a range from 0 to 12 minutes.
Sarcopenia | 6 months
  Geriatric multidimensional assessment for the evaluation of Sarcopenia by SARC-f questionnaire in patients over 65 years old. Score Range 0-10 points.
Assessment of endothelial function | 6 months
  Evaluation of endothelial function by Digital semiplethysmographic method through EndoPAT
Pulse Wave velocity assessment | 6 months
  Evaluation of carotid-femoral pulse wave velocity by SphygmoCor
Determination of lipopolysaccharide | 6 months
  Evaluation of lipopolysaccharide by ELISA sandwich

SECONDARY OUTCOMES:
Study of functional gut microbiota | 6 months
  Evaluation of gut microbiota by omics methods
Evaluation of gut microbiota | 6 months
  Evaluation of gut microbiota by bioinformatic methods
Evaluation of platelets activation | 6 months
  Evaluation of platelets activation biomarkers by ELISA sandwich method
Evaluation of oxidative stress | 6 months
  Evaluation of oxidative stress biomarkers by ELISA sandwich method
Evaluation of inflammatory cytokines | 6 months
  Evaluation of inflammatory cytokines (Interleukine-6, Interleukine-1) by ELISA sandwich method
Evaluation of endocan levels | 6 months
  Evaluation of values of endocan by ELISA sandwich method
Evaluation of hepcidin | 6 months
  Evaluation of circulating levels of hepcidin by ELISA sandwich method
Determination of mammalian target of rapamycin (mTOR) | 6 months
  Evaluation of mTOR by ELISA sandwich method
Proteomic analysis | 6 months
  Proteomics evaluation for study of post-translational modifications of circulating protein by reference Peptides markers

CONTACTS AND LOCATIONS:
Overall Officials: Angela Sciacqua, MD, Principal Investigator — University of Catanzaro
Locations (1):
- University Magna Graecia Mater Domini Hospital, Catanzaro, Calabria, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Correale M, Paolillo S, Mercurio V, Limongelli G, Barilla F, Ruocco G, Palazzuoli A, Scrutinio D, Lagioia R, Lombardi C, Lupi L, Magri D, Masarone D, Pacileo G, Scicchitano P, Matteo Ciccone M, Parati G, Tocchetti CG, Nodari S. Comorbidities in chronic heart failure: An update from Italian Society of Cardiology (SIC) Working Group on Heart Failure. Eur J Intern Med. 2020 Jan;71:23-31. doi: 10.1016/j.ejim.2019.10.008. Epub 2019 Nov 8. PMID 31708358
- [Background] Tomasoni D, Adamo M, Anker MS, von Haehling S, Coats AJS, Metra M. Heart failure in the last year: progress and perspective. ESC Heart Fail. 2020 Dec;7(6):3505-3530. doi: 10.1002/ehf2.13124. Epub 2020 Dec 5. PMID 33277825
- [Background] Gentlesk PJ, Sauer WH, Gerstenfeld EP, Lin D, Dixit S, Zado E, Callans D, Marchlinski FE. Reversal of left ventricular dysfunction following ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2007 Jan;18(1):9-14. doi: 10.1111/j.1540-8167.2006.00653.x. Epub 2006 Nov 1. PMID 17081210
- [Background] Parati G, Lombardi C, Castagna F, Mattaliano P, Filardi PP, Agostoni P; Italian Society of Cardiology (SIC) Working Group on Heart Failure members. Heart failure and sleep disorders. Nat Rev Cardiol. 2016 Jul;13(7):389-403. doi: 10.1038/nrcardio.2016.71. Epub 2016 May 12. PMID 27173772